CLINICAL TRIAL: NCT00343668
Title: A Phase II Study of S-1 and Irinotecan Combination Chemotherapy in Patients With Advanced Gastric Cancer as a First-Line Therapy
Brief Title: S-1 and Irinotecan Combination Chemotherapy for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Cancer Study Group (Other)
Responsible Party: Baek-Yeol Ryoo, Korea Cancer Center Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-ST05-02
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2006-06

CONDITIONS: Gastric Cancer
Keywords: advanced gastric cancer; First-line therapy; S-1; irinotecan
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: S-1, irinotecan — S-1, 40 mg/m2 PO twice daily, days 1-14 irinotecan, 150 mg/m2 IV, day 1

SUMMARY:
The primary goal of this phase II trial is to evaluate the response rate of combination chemotherapy with S-1 and Irinotecan in patients with advanced gastric cancer as a first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven unresectable adenocarcinoma of stomach
* With uni-dimensionally measurable disease (at least longest diameter 2 cm on conventional CT scan, x-ray or physical examination, or 1cm on spiral CT scan)
* Age 18 to 70 years old
* Estimated life expectancy of more than 3 months
* ECOG performance status of 2 or lower
* Adequate bone marrow function(absolute neutrophil count [ANC] ≥1,500/µL, hemoglobin ≥9.0 g/dL,and platelets ≥100,000/µL)
* Adequate kidney function (serum creatinine < 1.5 mg/dL)
* Adequate liver function (serum total bilirubin < 2 times the upper normal limit (UNL); serum transaminases levels <3 times [<5 times for patients with liver metastasis] UNL)
* No prior chemotherapy but prior adjuvant chemotherapy finished at least 6 months before enrollment was allowed. (but, prior adjuvant chemotherapy with capecitabine or S-1 or camptothecin analogues was excluded)
* No prior radiation therapy for at least 4 weeks before enrollment in the study

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Central nervous system (CNS) metastases or prior radiation for CNS metastases
* Gastric outlet obstruction or intestinal obstruction
* Evidence of gastrointestinal bleeding
* The patient has bony lesions as the sole evaluable disease.
* Past or concurrent history of neoplasm other than stomach cancer, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions

  * Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
  * History of significant neurologic or psychiatric disorders including dementia or seizures
  * Active uncontrolled infection
  * Other serious underlying medical conditions which could impair the ability of the patient to participate in the study
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy
* concomitant drug medication; The following drugs cause drug interaction with S-1.

  i. Warfarin, phenprocoumon: increase bleeding tendency ii. Increase blood concentration of phenytoin iii. sorivudine: inhibit DPD -> increase toxicity according to fluoropyrimidine iv. allopurinol : decrease activity of S-1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
response rate | best response

SECONDARY OUTCOMES:
treatment-related toxicities | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Baek-Yeol Ryoo, M.D., Ph.D., Principal Investigator — Korea Institute of Radiological and Medical Sciences
Locations (7):
- South Korea (7):
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeolanam-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Inha University hospital, Inchon
  - Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul
  - Yonsei Cancer Center, Seoul
  - Seoul Veterans Hospital, Seoul
  - Korea Institute of radiological and Medical Sciences, Seoul